CLINICAL TRIAL: NCT03040648
Title: Detection of Intravascular Penetration During Cervical Transforaminal Epidural Block: a Comparison of Digital Subtraction Angiography and Real Time Fluoroscopy
Brief Title: Detection of Intravascular Penetration During Cervical Transforaminal Epidural Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Younghoon Jeon, Professor, Kyungpook National University Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KNUH 2016-05-039-001
Record Dates: First submitted 2017-01-29; First posted 2017-02-02 (Estimated); Last update posted 2017-02-02 (Estimated); Status verified 2017-01

CONDITIONS: Diagnostic Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cervical TFEB under DSA (Experimental): cervical TFEB was performed under DSA
  Interventions: Device: DSA
- TFEB under RTF (Active Comparator): cervical TFEB was performed under RTF
  Interventions: Device: RTF

INTERVENTIONS:
Device: DSA — DSA was used for detection of intravascular injection
  Arms: cervical TFEB under DSA
Device: RTF — RTF was used for detection of intravascular injection
  Arms: TFEB under RTF

SUMMARY:
Transforaminal epidural block (TFEB) with local anesthetics and steroid is effective to treat spinal radicular pain. However, inadvertent intravascular injection can lead to severe neurologic complications. Digital subtraction angiography (DSA) during epidural block might increase the detection rate of intravascular penetration, compared to real-time fluoroscopy (RTF). But, DSA has disadvantages, such as additional radiation exposure to physicians and participants and the high cost of the new and upgraded fluoroscopic equipment. In this study, it was designed to compare DSA and RTF for detection of intravascular penetration in the same participant who underwent cervical TFEB.

The investigators prospectively examined the participants who received cervical TFEB. The needle position was confirmed using biplanar fluoroscopy and 2 ml of nonionic contrast media was injected at the rate of 0.5 ml/sec under RTF. Thirty seconds later, 2 ml of nonionic contrast media was injected at the rate of 0.5 ml/sec under DSA.

ELIGIBILITY:
Inclusion Criteria:

* participants with radiating pain from spinal stenosis and herniated nucleus pulposus.

Exclusion Criteria:

* pregnancy, allergic to contrast media, participants refusal, and participants with persistent contraindication to nerve block such as coagulopathy and infection of the injection site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence of intravascular injection | 4 seconds after injection of contrast media
  The incidence of intravascular injection during cervical transforaminal block

CONTACTS AND LOCATIONS:
Overall Officials: Saeyoung Kim, MD, Study Chair — Kyungpook National University Hospital
Locations (1):
- Kyungpook National University Hospital, Daegu, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jeon Y, Kim S. Detection of Intravascular Injection During Cervical Transforaminal Epidural Injection: A Comparison of Digital Subtraction Angiography and Real Time Fluoroscopy. Pain Physician. 2018 Mar;21(2):E181-E186. PMID 29565961